CLINICAL TRIAL: NCT07041385
Title: Comparing the Efficacy of 75mg Versus 150mg Aspirin for the Prevention of Preeclampsia in High-Risk Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalamar Hospital (Other)
Responsible Party: Principal Investigator, Hafiz Wajahat Naseem, Post Graduate Resident in Gynae and OBS. Department, Shalamar Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB - 830
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia (PE)
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A: 75 mg aspirin nightly.
  Interventions: Drug: Aspirin 75 mg
- Group B (Experimental): Group B: 150 mg aspirin nightly.
  Interventions: Drug: Aspirin 150 mg

INTERVENTIONS:
Drug: Aspirin 75 mg — This study aims to evaluate the effectiveness of 75 mg aspirin versus 150 mg aspirin in preventing preeclampsia among individuals with high risk for the condition.
  Eligible women attending the antenatal clinic were screened by history, physical exam, and uterine artery Doppler. Risk assessment was entered into the Fetal Medicine Foundation software. Participants were randomized:
  Group A: 75 mg aspirin nightly. Group B: 150 mg aspirin nightly.
  Arms: Group A
Drug: Aspirin 150 mg — This study aims to evaluate the effectiveness of 75 mg aspirin versus 150 mg aspirin in preventing preeclampsia among individuals with high risk for the condition.
  Eligible women attending the antenatal clinic were screened by history, physical exam, and uterine artery Doppler. Risk assessment was entered into the Fetal Medicine Foundation software. Participants were randomized:
  Group A: 75 mg aspirin nightly. Group B: 150 mg aspirin nightly.
  Arms: Group B

SUMMARY:
This study aims to evaluate the effectiveness of 75 mg aspirin versus 150 mg aspirin in preventing preeclampsia among individuals with high risk for the condition. Existing literature suggests that the 150 mg aspirin dose may exhibit superior efficacy, yet inconclusive evidence exists in our local setting.

DETAILED DESCRIPTION:
Pre-eclampsia is a major factor in both maternal and fetal morbidity and mortality. The most widely investigated preeclampsia prevention medication is low dose Aspirin. However, guidelines differ considerably regarding the prophylactic dose of Aspirin for preeclampsia. Pre-eclampsia (PE) affects 5-7% of all pregnancies and along with eclampsia is the major contributor to maternal morbidity and 10-15% of maternal mortality and also perinatal mortality. Low dose aspirin administration can reduce vasoconstriction and decreases thrombosis of the vessels related to placenta, thereby increases blood flow and protects against to pregnancy related complication like preeclampsia, IUGR or FGR. One of the major therapeutic interventions to prevent preeclampsia is the use of Aspirin (a COX-II inhibitor with anti-inflammatory and anti-thrombotic properties). Initiating low-dose aspirin (LDA) therapy in early pregnancy from 12 weeks can prevent the onset of pre-eclampsia or delay it. The antiplatelet and vasodilatory effect of aspirin induced by the inhibition of cyclooxygenase-1 (COX-1) and reduced production of thromboxane, a potent vasoconstrictor and platelet aggregator, enhances placental blood circulation. Moreover, potential anti-inflammatory properties can improve endothelial dysfunction and oxidative stress, which are the central pieces of preeclampsia mechanisms.

The dose of aspirin used in most hospital settings is low dose, which has its benefits outweigh the risks and side effects of the drug. Many studies evaluated low doses of Aspirin 60-80mg showing a 10%-50% reduction in the incidence of preeclampsia, while a few studies also evaluated the efficacy of a 150mg dose. To our knowledge, this is among very few studies to investigate the effectiveness of relatively higher doses of aspirin in the Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

1. Screen positive women
2. Age 18 - 30 y
3. Gestational Age 11 - 13+6 weeks
4. Singleton Pregnancy
5. Estimated risk for preterm PE of > 1 in 100 (Reference - Fetal Medicine Foundation)

Exclusion Criteria:

1. Screen negative women
2. Age > 30 y
3. Gestational Age > 14 weeks
4. Multiple Gestation
5. Estimated risk for preterm PE of < 1 in 100 (Reference - Fetal Medicine Foundation)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All Pregnant Females
Enrollment: 340 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pre - eclampsia | 9 months
  PE (Pre-eclampsia) Yes / No Early Onset - Pre-eclampsia (<34 weeks) Yes / No Late Onset - Pre-eclampsia (>34 weeks) Yes / No

SECONDARY OUTCOMES:
Delivery | 9 months
  Preterm - Pre-eclampsia Delivery (<37 weeks) Yes / No Term Delivery - Pre-eclampsia (>37 weeks) Yes / No

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations the data will be placed in password protected laptop ,only Principal investigator can access the data.